CLINICAL TRIAL: NCT02559154
Title: An Open-Label Phase IV Study of the Efficacy of Bortezomib-based Combination Therapy the Treatment of Subjects With Multiple Myeloma
Brief Title: Modified Bortezomib-based Combination Therapy for Multiple Myeloma
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Daolin Wei, Principal Investigator,Doctor, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2010K059
Record Dates: First submitted 2015-09-21; First posted 2015-09-24 (Estimated); Last update posted 2018-05-04 (Actual); Status verified 2018-05

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib; Dexamethasone; Doxorubicin; Cyclophosphamide; Thalidomide

ARMS (2):
- modified BZ group (Experimental): Patients with newly diagnosed or pre-treated MM(prior therapy not including bortezomib) received regimen with bortezomib (1.6mg/㎡) as an intravenous bolus once weekly on day 1, 8 in a 3 weeks cycle, in combination with dexamethasone,with or without doxorubicin/ cyclophosphamide/mitoxsnteone/thalidomide
  Interventions: Drug: Bortezomib; Drug: Dexamethasone; Drug: Doxorubicin; Drug: Cyclophosphamide; Drug: Mitoxsnteone; Drug: Thalidomide
- conventional BZ group (Active Comparator): Patients with newly diagnosed or pre-treated MM(prior therapy not including bortezomib) received bortezomib (1.3mg/㎡) administration twice weekly on day 1,4, 8,11 in a 3 weeks cycle, in combination with dexamethasone,with or without doxorubicin/ cyclophosphamide/mitoxsnteone/thalidomide
  Interventions: Drug: Bortezomib; Drug: Dexamethasone; Drug: Doxorubicin; Drug: Cyclophosphamide; Drug: Mitoxsnteone; Drug: Thalidomide

INTERVENTIONS:
Drug: Bortezomib
  Other Names: velcade
Drug: Dexamethasone
Drug: Doxorubicin
Drug: Cyclophosphamide
Drug: Mitoxsnteone
Drug: Thalidomide

SUMMARY:
To investigate the efficacy of a modified bortezomib based combination therapy for patients with multiple myeloma.

DETAILED DESCRIPTION:
Multiple myeloma (MM) is a common hematological malignancy in Chinese elderly population. The application of novel drugs improved the clinical outcome and survival of MM patients,even though MM remains an incurable hematological malignancy. Bortezomib is a typical one among these novel agents, its application resulted in great success, but its adverse events and high expense restricted its widely usage. Investigators modified the dose and frequency of bortezomib administration in combination therapy: Patients in the modified group received regimen with bortezomib (1.6mg/㎡) as an intravenous bolus once weekly on day 1, 8 in a 3 weeks cycle, in combination with dexamethasone,with or without doxorubicin/ cyclophosphamide/mitoxsnteone/thalidomide，while patients in the control group received similar combination therapy except with conventional bortezomib (1.3mg/㎡) administration twice weekly on day 1,4, 8,11.

The aim of this study is to investigate whether the modified bortezomib-based therapy may attain a similar efficacy as the conventional ones.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of multiple myeloma based on standard diagnosis criteria:

  * plasmacytomas on tissue biopsy
  * bone marrow plasmacytosis
  * monoclonal immunoglobulin spike on serum electrophoresis
  * lytic bone lesions.
* Must have relapsed or relapsed/refractory disease
* 18 years of age or older
* All baseline studies must be performed within 21 days of enrollment.
* ECOG performance status of 0 to 2

Exclusion Criteria:

* Renal insufficiency (serum creatinine levels > 2mg/dL)
* Concomitant therapy medications that include corticosteroids
* Peripheral neuropathy of Grade 3 or greater or painful Grade 2
* Evidence of mucosal or internal bleeding and/or platelet refractory
* ANC < 1000 cells/mm3
* Hemoglobin < 8.0 g/dL
* AST (SGOT and ALT) > 2 x ULN
* Intolerance to bortezomib or CC-5013 in the past or significant allergy to either compound, boron or mannitol
* Known hypersensitivity to thalidomide or the development of erythema nodosum
* Active infection or serious co-morbid medical condition
* Pregnant or breast-feeding women
* Prior malignancy with the last three years except adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, in situ breast cancer, on in-situ prostate cancer

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2010-07; Primary Completion 2018-10 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
disease responses to treatment | one year
  Response evaluated by changes of serum M-component(g/L) through Serum quantitative immunoglobulins and Serum immunofixation electrophoresis.
  (g/L)

CONTACTS AND LOCATIONS:
Overall Officials: Guohua Liu, MD, Study Chair — Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Shanghai General Hospital, Shanghai, China